CLINICAL TRIAL: NCT04582305
Title: Intralesional Bleomycin Treatment of Keloids Using an Electronic Pneumatic Jet Injector: a Double-blind Randomized, Placebo-controlled Trial With Split-lesion Design
Brief Title: Bleomycin Jet Injections in Keloids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Principal Investigator, M.B.A. van Doorn, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLEO JET
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Keloid
Keywords: Keloid; Dermatology; Bleomycin; Jet-injection
MeSH Terms: conditions — Keloid | interventions — Bleomycin; Saline Solution

STUDY DESIGN:
Intervention Model Description: A single center, double-blind (patient and investigator), randomized, placebo-controlled study with a split-lesion design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bleomycin jet-injections (Active Comparator): This study consists of a split-lesion design in which the keloid scar will receive three consecutive treatments with an interval of 4 weeks of: 1) bleomycin and 2) placebo (NaCl 0,9%), administered with an electronic pneumatic jet injector. A single injection of 100 μL will be given per 1 cm2, with a maximum of 20 injections per treatment. The maximum dosage of bleomycin per treatment will be 2 mL, corresponding to 2 USP-E (units) of bleomycin. The maximum cumulative dosage of bleomycin will be 6 USP-E in this study.
  Interventions: Drug: Bleomycin
- Placebo jet-injections (Placebo Comparator): This study consists of a split-lesion design in which the keloid scar will receive three consecutive treatments with an interval of 4 weeks of: 1) bleomycin and 2) placebo (NaCl 0,9%), administered with an electronic pneumatic jet injector. A single injection of 100 μL will be given per 1 cm2, with a maximum of 20 injections per treatment. The maximum dosage of normal saline per treatment will be 2 mL.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Bleomycin — Intralesional bleomycin treatment administered with an electronic pneumatic jet injector
  Arms: Bleomycin jet-injections
Drug: Normal saline — Intralesional placebo treatment of normal saline administered with an electronic pneumatic jet injector
  Arms: Placebo jet-injections

SUMMARY:
This is a single center, double-blind (patient and investigator), randomized, placebo-controlled study with a split-lesion design, in which selected keloids will receive three consecutive treatments of a) bleomycin and b) placebo (saline (NaCl 0,9%)), administered with an electronic pneumatic jet injector.

DETAILED DESCRIPTION:
This is a single center, double-blind (patient and investigator), randomized, placebo-controlled study with a split-lesion design.All study procedures will be performed at the Department of Dermatology, Erasmus MC Medical Center in patients referred for scar treatment to our outpatient clinic.

Clinical photos will be obtained after signing the informed consent form by patient and investigator. Study visits and clinical assessments will be scheduled at baseline, 4 weeks, 8 weeks, and 12 weeks. Measurements include clinical photography, scar volume measured by 3D-camera, POSAS questionnaire, laser speckle contrast imaging to visualize keloid scar vascularization, measurement of residue formation on the skin, and a treatment related questionnaire. The keloid will be divided into two treatment areas, and randomly assigned to three consecutive treatments of: a) bleomycin and b) placebo (saline (NaCl 0,9%)), administered with an electronic pneumatic jet injector.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent;
2. Subject is ≥ 18 years of age at time of screening;
3. Subject has at least one keloid scar of ≥ 4 cm in length, or two separate keloids with a length of ≥2cm, with a minimum > 1.0 cm apart in the same anatomical region.
4. Subject is willing to fill in questionnaires and take photos using an e-diary application on their phone.

Exclusion Criteria:

1. Known hypersensitivity to any component of the test materials;
2. Pregnant or breast-feeding women (pregnancy test prior to treatment);
3. Previous bleomycin treatment of the keloid within the last 12 weeks prior to screening.
4. Non-response to previous bleomycin treatments of the keloid.
5. Any medical or psychiatric condition which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-11-18 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Volume reduction | 12 weeks
  Volume reduction of scar tissue in mm^3.

SECONDARY OUTCOMES:
Clinical efficacy using Patient and Observer Scar Assessment Scale (POSAS) | 12 weeks
  Evaluation of clinical efficacy using Patient and Observer Scar Assessment Scale. The POSAS consists of six items (vascularization, pigmentation, thickness, relief, pliability and surface). Each item will be scored on a scale from 1 (normal skin) to 10 (worst scar). The scores of these six items result in the 'POSAS total score', also on a scale from 1 (normal skin) to 10 (worst scar).
Vascular perfusion | 12 weeks
  Evaluation of changes in keloid vascular perfusion using Laser Speckle Contrast Imaging.
Residue formation on skin | 30 minutes
  Evaluation of the average residue formation on skin in percentage of the injection volume.
Procedure related pain | 30 minutes
  Evaluation of the procedure related pain using a numerical rating scale (NRS) score. This scale ranges from 0-10 points, with higher scores indicating greater pain intensity.
Local skin reactions | 12 weeks
  Evaluation of the local skin reactions using self-taken photos in an e-diary.
Treatment satisfaction | 12 weeks
  Evaluation of treatment satisfaction using a 5-point Likert scale. This scale ranges from -2 to 2 points, with higher scores indicating higher satisfaction.
Incidence of Treatment-Emergent Adverse events [Safety and Tolerability]. | 12 weeks
  Evaluation of safety and tolerability by evaluating all adverse events. Patients will daily be asked to take pictures of the treated lesion(s), and to report any adverse event via an digital e-diary application.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn van Doorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Eramsus Medical Centre, Dermatology department, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No